CLINICAL TRIAL: NCT06513429
Title: Clinical Study on Evaluating the Efficacy and Safety of IM19 CAR-T Cell Therapy in Patients With Refractory Systemic Lupus Erythematosus
Brief Title: IM19 CAR-T Cell Therapy in Refractory Systemic Lupus Erythematosus (SLE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Mu Rong, Chief of Department of Rheumatology and Immunology, Peking University Third Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM19SLE01
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Refractory Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; CAR-T cell
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T cell therapy group (Experimental): Administration of IM19 CAR-T cells at a dose of 1×10^6/kg CAR-T cells for patients 1 to 3, and 1×10^8 CAR-T cells for patient 4 to 6.
  Interventions: Biological: IM19 CAR-T cells

INTERVENTIONS:
Biological: IM19 CAR-T cells — IM19 CAR-T cells by intravenous infusion.
  Other Names: CD19 CAR-T cells

SUMMARY:
The study is a single-arm, open-label clinical trial intended to recruit 6 refractory SLE subjects who meet the inclusion and exclusion criteria. The subjects will receive IM19 CAR-T cell infusion therapy at a dose of 1×10^6/kg or 1×10^8 CAR-T cells . The primary endpoint is to evaluate the improvement in SLE disease activity (SLEDAI-2K) at 90 days and the occurrence of adverse events related to IM19 CAR-T cell infusion within 28 days post-infusion. Additionally, the long-term efficacy was evaluated, including the improvement of SLEDAI-2K score and achieving lupus low disease activity (LLDAS) at day 180 and day 360, and renal response at day 180 and day 360. The persistence and duration of IM19 CAR-T cells in the peripheral blood of subjects will also be evaluated. The study plan includes five phases: screening phase, cell collection phase, lymphodepletion pretreatment phase, cell infusion phase, and follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* 1)The subject was diagnosed with systemic lupus erythematosus and met the classification criteria of EULAR/ACR 2019 SLE (see Annex 2)
* 2) Age ≥ 18 years old, ≤ 65 years old
* 3) Weight ≥ 40 kg
* 4) Meets the current clinical standards for refractory systemic lupus erythematosus: the disease remains active or relapses and progresses after systemic treatment using the current standard treatment regimen, including steroids (sufficient or shock therapy), immunosuppressants (cyclophosphamide or mycophenolate mofetil), and biologics (belizumab or Rituximab)
* 5) Currently, one or more of the following stable dose standard therapies are being used to treat SLE: steroids, antimalarial drugs, immunosuppressants. If the subject is receiving steroids, the following conditions must be met: at screening time and during screening period, the maximum dose of steroids is 30mg/day prednisone (or equivalent dose). Before screening, the dose of steroids should remain stable for ≥ 7 days. During the screening period, the dose of steroids adjustment should not exceed 5mg/day prednisone (or equivalent dose). If the subject is receiving treatment with antimalarial drugs and/or conventional immunosuppressants: the start time of drug treatment must be ≥ 12 weeks before screening. Maintain a stable dose of medication for at least 8 weeks before and during screening. Before the screening period, if biological agents (such as belizumab or Telitacicept) are used, they need to be discontinued for at least 4 weeks before screening.
* 6) Disease activity score (SLEDAI-2K) with a score of 10 or above (refer to Attachment 3)
* 7) Women of childbearing age who tested negative for blood pregnancy before the start of the trial and agreed to take effective contraceptive measures during the trial period until the last follow-up
* 8) Male participants whose partners have fertility agree to take effective contraceptive measures during the trial period until the last follow-up

  * 9) Those who voluntarily participate in this experiment and sign an informed consent form.

Exclusion Criteria:

* 1) After evaluation by researchers, it is determined that the subject has diseases that are not suitable for participation in this study, such as life-threatening conditions (e.g., catastrophic antiphospholipid syndrome, acute severe renal failure, acute severe central nervous system disease manifestations).
* 2) The research subject has a history of alcohol or drug abuse within the past 24 weeks.
* 3) The research subject has a history of malignant tumors other than B-cell lymphoma.
* 4) Major surgery (including joint surgery) was performed within 24 weeks prior to screening, or surgery is planned within 24 weeks after enrollment in the study.
* 5) The research subject has overlapping mixed connective tissue diseases and other syndromes that affect the judgment of disease activity.
* 6) The research subject has human immunodeficiency virus (HIV) infection, selective IgA deficiency, T-cell deficiency virus infection, chronic hepatitis B or C virus infection, or SARS-CoV-2 [severe acute respiratory syndrome coronavirus 2] infections.
* 7) The research subject has a known active tuberculosis (TB) infection or bacterial infection.
* 8) History of myocardial infarction, cardiac angioplasty or stent placement, unstable angina, active arrhythmia, or other clinically significant heart disease within 6 months prior to screening initiation.
* 9) History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to screening initiation.
* 10) The research subject's alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) levels are ≥3×ULN, or bilirubin >1.5×ULN, excluding laboratory test abnormalities due to SLE hepatitis.
* 11) The research subject has stage 4 chronic kidney failure, indicated by an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m², or serum creatinine >2.5 mg/dL. During the screening visit (V1), the research subject presents with any of the following significant hematological abnormalities: a. Hemoglobin <7.0 g/dL b. CD4+ T lymphocytes <200/mm³ c. Absolute neutrophil count <500/mm³ d. CD4+ T lymphocytes <500/mm³ with a neutrophil count <1000/mm³ e. Platelets <25,000/mm³.
* 12) Treatment with CD20 monoclonal antibodies was used within the past 6 months.
* 13) Conditions that the researcher considers unsuitable for inclusion in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of SLEDAI-2K score at 90 days after IM19 CAR T cell transfusion. | 90 days
  Change from baseline of SLEDAI-2K score at 90 days after IM19 CAR T cell transfusion. Range [0,105], higher values indicate worse disease activity.
Adverse events related to IM19 CAR-T cell therapy within 28 post-infusion. | 90 days
  The occurrence of adverse events related to IM19 CAR-T cell therapy within 28 post-infusion.

SECONDARY OUTCOMES:
Change from baseline of SLEDAI-2K score at day 180 and day 360 after IM19 CAR T cell transfusion. | 180 days and 360 days
  Change from baseline of SLEDAI-2K score at day 180 and day 360 after IM19 CAR T cell transfusion. Range [0,105], higher values indicate worse disease activity.
Achieving low disease activity status (LLDAS) at day 180 and day 360 post IM19 CAR-T cell infusion. | 180 and 360 days
  Achieving low disease activity status (LLDAS) at day 180 and day 360 post IM19 CAR-T cell infusion.
Renal response at day 180 and day 360 post CAR-T cells infusion. | 180 and 360 days.
  Complete renal response was defined as 24-hour urine protein ≤0.5 g/day; partial renal response was defined as proteinuria ≥50% reduction from baseline and 24-hour proteinuria <3.5 g/day or protein-creatinine ratio (PCR) <3.0mg/g, with stable or improved kidney function (±10%-15% of baseline).
The persistence and duration of IM19 CAR-T cells in the peripheral blood of subjects. | 360 days
  The persistence and duration of IM19 CAR-T cells in the peripheral blood of subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Universitiy Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No